CLINICAL TRIAL: NCT07140809
Title: a Multiple-center, Randomized, Double-blind, Placebo-controlled, Multiple-dose Escalation Phase Ib/Ⅱa Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetic Characteristics of JMT202 Injection in Chinese Participants With Hypertriglyceridemia
Brief Title: a Phase 1b/2a Study of JMT202 Injection in Participants With Hypertriglyceridemia
Acronym: phase Ib/Ⅱa st
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JMT202-002
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMT202 (Experimental): Participants received JMT202 as an injection according to the protocol.
  Interventions: Biological: JMT202 injection
- Placebo (Placebo Comparator): Participants received placebo as an injection according to the protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: JMT202 injection — Subcutaneous injection
  Arms: JMT202
Other: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of multiple subcutaneous injections of JMT202 injection in Chinese participants with hypertriglyceridemia

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years old (at the time of signing the informed consent form), gender not limited.
* The weight is ≥45.0 kg (for females) or ≥50.0 kg (for males), and the body mass index is between 24.0 and 40.0 kg/m ² (including the cut-off value). The body mass index is calculated as [BMI= weight (kg)/height 2 (m ²)].
* TG>300 mg/dL (3.39 mmol/L) within 28 days before screening; During the screening period, the TG of the participants met the following requirements: ① Two TG values within the screening period, with an interval of ≥7 days, and both TG values met the requirement of 300 mg/dL≤TG<1000 mg/dL (11.30 mmol/L); ② The last TG test was less than 7 days before administration (D1).
* Participants need to meet:

  1. Receive stable lipid-lowering treatment for ≥28 days before screening;
  2. Accept lipid-lowering medications before screening of less than 28 days, but random stable lipid-lowering therapy, 28 days or more before test TG and D - 1 > 300 mg/dL (the tendency for 3.39 L) screening of unused lipid-lowering within 28 days before,
  3. During the screening period, at least one screening should be conducted at a concentration of 300 mg/dL (3.39 mmol/L) ≤TG<500 mg/dL (5.65 mmol/L).
  4. Screening unused lipid-lowering, within 28 days before screening period two TG 500 mg/dL or higher tendency (5.65 L), need before random stable lipid-lowering therapy, 28 days or TG test and D - 1 > 300 mg/dL (the tendency for 3.39 L).Lipid-lowering treatment: niacin ≥375 mg/ day, prescription fish oil, fibrates, statins, ezetimibe, etc. PCSK9 inhibitors need to be stable for 6 months before screening.
* Some participants (at least 4 cases per dose group) had MRI-PDFF≥8%;
* From 28 days before screening to the entire trial period, participants should maintain their original diet, exercise and lifestyle habits as much as possible, and avoid alcohol and strenuous exercise within 48 hours before each visit.
* Participants and their partners agree that they must use effective and reliable contraceptive methods from the signing of the informed consent form until 6 months after the end of the trial (female participants are not allowed to use hormonal contraceptives from 14 days before screening until the entire trial period) to prevent pregnancy in either female or male participants' partners. Male participants had no sperm donation plans from signing the informed consent form to 6 months after the end of the trial, and female participants had no egg donation plans from signing the informed consent form to 6 months after the end of the trial.
* Participants voluntarily join the clinical trial and sign the informed consent form, and have the ability to communicate normally with the researchers while abiding by the trial requirements.

Exclusion Criteria:

* Weight changed by ≥5% within the 3 months prior to randomization, or who planned to lose weight throughout the trial period;
* Screening products targeting the FGF21 target that have been used within the previous year, such as BIO89-100, DR10624, etc.
* Participants with Type 1 diabetes No stable hypoglycemic drug treatment within 3 months prior to screening or randomization (the use of glucagon-like peptide-1 receptor agonists, single-target or multi-target drugs, thiazolidinediones or insulin was prohibited from 3 months prior to screening until the entire trial period) Other oral or injectable drugs should have been stably treated for ≥3 months before screening and the dose should be maintained stably throughout the trial period, or the glycated hemoglobin should be ≥9.5% during the screening period.
* Participants who are known or suspected of having familial hyperchylomicemia, lipoprotein lipase injury or deficiency (Fredrickson type 1), apolipoprotein C-II deficiency or familial lipoprotein dyslipidemia (Fredrickson type 3);
* Participants with a history of gallbladder disease and have symptoms before Screen or randomly (such as common bile duct stones, multiple gallbladder stones, etc., unless the gallbladder has been removed and the removal time is ≥6 months);
* Participants had a history of acute pancreatitis attacks or chronic pancreatitis within 12 months prior to screening or randomization;
* Subjects with atherosclerotic cardiovascular diseases in the 6 months prior to screening or randomization, including acute coronary syndrome, stable coronary heart disease, post-revascularization, ischemic cardiomyopathy, ischemic stroke, transient ischemic attack, peripheral atherosclerotic disease, etc., or those diagnosed with a high risk of atherosclerotic cardiovascular disease;
* There were major cardiovascular and cerebrovascular diseases in the 6 months prior to screening or randomization;
* Having a history of malignant tumors in the past five years (excluding cured basal cell carcinoma of the skin, localized squamous cell carcinoma of the skin or carcinoma in situ of cervical cancer), or potential malignant tumors currently under assessment;
* Participants have experienced severe infections within the three months prior to screening, including but not limited to: severe pneumonia, lung abscess, meningitis, cellulitis, etc., and are judged by the researchers as unsuitable to participate in this trial;
* Participants with poor blood pressure control during the screening period (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg); Or the antihypertensive drugs of the participants have not been stable for ≥3 months before screening or randomization (thiazide diuretics and beta-blockers are prohibited from 3 months before screening to the entire trial period).
* Participants test positive for any one of hepatitis B surface antigen, hepatitis C virus antibody, Treponema pallidum antibody or human immunodeficiency virus antibody;
* Other lipid regulators (excluding lipid-lowering drugs in inclusion criterion 4) were used from 28 days before screening/randomization to the entire trial period (≥3 days), including niacin (<375 mg/ day), over-the-counter or non-pharmaceutical strength fish oil, red rice yeast supplements, garlic supplements, soy isoflavone supplements, sterols/sterol products, polyphenols, etc.
* In the opinion of the investigator, the participants have symptoms such as dermatitis or abnormal skin around the abdominal administration site;
* Participants with a history of severe drug or food allergies, who have used immunosuppressant drugs, or who are determined by the researcher to be allergic to the investigational drug;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of TEAE | Day 1 to 99
Number of participants with vital sign abnormalities | Day 1 to 99
Number of participants with physical examination abnormalities | Day 1 to 99
Number of participants with laboratory tests abnormalities | Day 1 to 99
Number of participants with 12-lead electrocardiogram abnormalities | Day 1 to 99
Number of participants with injection site reactions abnormalities | Day 1 to 63

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Peking University, Beijing, Beijing Municipality, China